CLINICAL TRIAL: NCT07201662
Title: Role of Empathy in the Links Between Binge Eating Disorder and Interpersonal Difficulties in the Context of Obesity in a Clinical Population
Brief Title: The Role of Empathy in the Links Between Binge Eating Disorder and Interpersonal Difficulties
Acronym: EMBED_OB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique de la Mitterie (Other)
Collaborators: Clinique les Peupliers (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-A00868-41; MR-P0010 (Other: National Agency for Safety and Medicines)
Record Dates: First submitted 2025-08-29; First posted 2025-10-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Obesity &Amp;Amp; Overweight
Keywords: obesity; binge eating disorder; Empathy
MeSH Terms: conditions — Obesity; Overweight; Binge-Eating Disorder | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Intervention Model Description: Single-center type 2 trial (interventional study with minimal risks and constraints)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Nutritional Rehabilitation (Experimental): Patients presenting for a "standard" stay, preparation for bariatric surgery, or post-surgical follow-up in the Nutritional Rehabilitation department
  Interventions: Other: Condensed and Revised Multifaceted Empathy Test; Other: Hospital Anxiety and Depression Scale; Other: Interpersonal Reactivity Index; Other: Vicarious Distress Questionnaire; Other: Binge Eating Scale

INTERVENTIONS:
Other: Condensed and Revised Multifaceted Empathy Test — Experimental emotional decoding task that measures the cognitive and affective dimensions of empathy based on performance (Edele et al., 2013; Grynberg et al., 2017).Participants view 40 photos of faces expressing either a positive or negative emotion and must identify the emotion (decoding) and then rate on a 1-9 scale the extent to which they share it (emotional sharing). The task lasts approximately 10 minutes on average.
Other: Hospital Anxiety and Depression Scale — A self-administered scale with 14 items, divided into two subscales of seven items, used to detect the presence of depression and anxiety. Non-cases or asymptomatic individuals (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
  The administration time is approximately 5 minutes.
Other: Interpersonal Reactivity Index — The Interpersonal Reactivity Index (Davis, 1980; Guttman & Laporte, 2002) is a 28-item self-report questionnaire measuring four dimensions of empathy: fantasy, perspective taking, empathic concern, and personal distress. Each item is rated on a 1-to-5 scale and provides a subscore for each dimension, with no overall total score. Administration takes approximately 5 minutes.
Other: Vicarious Distress Questionnaire — The Vicarious Distress Questionnaire (Grynberg et al., 2012) is an 18-item self-report scale assessing distress experienced in response to others' suffering and its impact on prosocial behaviors. It includes three dimensions-distress, support, and avoidance-each yielding a specific subscore. Administration takes approximately 5 minutes.
Other: Binge Eating Scale — The Binge Eating Scale (Gormally et al., 1982; Brunault et al., 2016) is a 16-item self-report questionnaire assessing the behavioral, emotional, and cognitive manifestations of binge eating disorder (BED) according to DSM-V criteria. The total score (0-46) reflects symptom severity and can be interpreted dimensionally or categorically (≥ 18 indicating significant symptomatology). Administration takes approximately 5 minutes.

SUMMARY:
Obesity, recognized as a chronic disease by the WHO since 1998, affects 22.1% of adults in the Hauts-de-France region. Beyond the physiological aspects, it is associated with psychological difficulties, particularly eating disorders such as binge eating disorder (BED), as well as interpersonal difficulties related to empathy. Empathy, which consists of cognitive (decoding emotion) and affective (sharing emotion) dimensions, appears to be reduced in obese adults compared to adults of normal weight. However, existing research remains limited and heterogeneous. It is therefore essential to explore the links between obesity, cognitive and affective empathy in greater detail, taking into account the role of BED, in order to better understand their impact on interpersonal relationships.

DETAILED DESCRIPTION:
Obesity has been recognized as a chronic disease by the World Health Organization since 1998. In the Hauts-de-France region, obesity affects 22.1% of adults.

Psychologically, it has been noted that obese individuals may experience intrapersonal difficulties (eating disorders such as binge eating disorder [BED], i.e., bulimia nervosa) and interpersonal difficulties, such as empathy disorders. Empathy is generally defined as a multidimensional concept, comprising two dimensions known as "cognitive" (decoding emotion) and "affective" (sharing emotion).

Empathic skills are significantly weaker in obese adults than in adults of normal weight. However, only ten studies were included in this research, and only two studies focused on affective empathy. In addition, the methodologies were highly heterogeneous (experimental tasks, self-assessment questionnaires). Therefore, the investigators believe it is essential to examine the links between obesity, cognitive empathy, and affective empathy in the adult population using a mixed methodology based on an experimental task and questionnaires. In addition, the investigators wish to examine the role of BED in explaining possible empathy disorders associated with obesity. Finally, the investigators wish to better understand the links between empathy difficulties and interpersonal difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* BMI ≥ 30 kg/m2
* French-speaking
* Enrolled in nutritional rehabilitation
* Written consent signed by the patient
* Affiliation with a social security system

Exclusion Criteria:

* Insufficient proficiency in the French language
* Minor patients, or patients under legal protection measures or deprived of liberty
* Lack of health insurance coverage
* Refusal to participate in the study
* Presence of neurological disorders
* Presence of cognitive disorders
* Presence of psychiatric disorders
* Presence of eating disorders such as anorexia or bulimia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
MET-Core | Enrollment
  Compare cognitive empathy skills obtained on the MET-Core between participants who are obese

SECONDARY OUTCOMES:
Empathy skills | Enrollment
  Compare the empathy skills self-reported by participants with obesity, based on the presence or absence of symptoms suggestive of BED.
Interpersonal difficulties assessed with the Inventory of Interpersonal Problems - Circumplex Scales (IIP-C) | Enrollment
  The IIP-C is a 64-item self-report questionnaire assessing interpersonal difficulties across eight sub-dimensions (each consisting of 8 items): Vindictive, Domineering, Intrusive, Overly Nurturant, Exploitable, Nonassertive, Socially Avoidant, and Cold.
  Each item is rated on a 5-point Likert scale (0 = not at all, 4 = extremely), reflecting the extent to which the statement represents a difficulty experienced by the participant in interpersonal relationships. For each sub-dimension, a mean score is computed, and a global score can also be calculated as the mean of all 64 items. Higher scores indicate greater interpersonal difficulties.
  The unit of measure will be the total IIP-C score (range: 0-4) and/or the subscale scores (range: 0-4). The average administration time is approximately 10 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique les Peupliers, Villeneuve-d'Ascq, France

IPD SHARING:
Plan to Share IPD: Undecided
No Plan Description for the moment